CLINICAL TRIAL: NCT02673489
Title: A Phase 3 Evaluation of Daclatasvir and Sofosbuvir With Ribavirin in Cirrhotic Subjects With Genotype 3 Chronic Hepatitis C Infection
Brief Title: A Study of Daclatasvir and Sofosbuvir With Ribavirin in Subjects With Cirrhosis and Genotype 3 Hepatitis C Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-379; 2015-004331-12 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daclatasvir (DCV) + Sofosbuvir (SOF) + Ribavirin (RBV) (Experimental): Oral dosing of DCV 60 mg tablet once daily + SOF 400 mg tablet once daily + RBV 1000-1200 mg tablet per day (weight based) for 24 weeks.
  Interventions: Drug: DCV; Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: DCV
Drug: SOF
Drug: RBV

SUMMARY:
The purpose of this study is to determine whether 24 weeks of Daclatasvir and Sofosbuvir with Ribavirin is safe and effective in the treatment of genotype 3 hepatitis C infected patients with liver cirrhosis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb (BMS) Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Genotype 3 HCV
* HCV RNA ≥10000 IU (International Unit)/mL
* Compensated Liver Cirrhosis
* BMI 18-40 kg/m2
* Previously treated for HCV or never treated for HCV

Exclusion Criteria:

* Infection with HCV other than Genotype 3. Mixed infection of any genotype
* Evidence of decompensated liver disease
* Previous exposure to NS5A inhibitors

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (12):
  - Keck Medical Center Of USC, Los Angeles, California
  - University Of California, San Francisco, San Francisco, California
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Ruth Rothstein Core Center, Chicago, Illinois
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc, Richmond, Virginia
- Canada (7):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Regina, Saskatchewan

REFERENCES:
- [Derived] Poordad F, Shiffman ML, Ghesquiere W, Wong A, Huhn GD, Wong F, Ramji A, Shafran SD, McPhee F, Yang R, Noviello S, Linaberry M; ALLY-3C study team. Daclatasvir and sofosbuvir with ribavirin for 24 weeks in chronic hepatitis C genotype-3-infected patients with cirrhosis: a Phase III study (ALLY-3C). Antivir Ther. 2019;24(1):35-44. doi: 10.3851/IMP3278. PMID 30382942
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 106 subjects enrolled, 78 participants entered the treatment period and received study treatment; 28 participants were enrolled but did not enter the treatment period. 26 were due to no longer meeting study criteria; 1 was due to poor/non-compliance (missed Day 1 visit); and 1 was other (missed screening window).
Groups:
- Treatment Naive: HCV treatment-naive: No previous exposure to any interferon (IFN) formulation (ie, IFN or peg-IFN), RBV, or any HCV DAAs
- Treatment Experienced: HCV treatment-experienced: Previous treatment with IFN/RBV, SOF + RBV, and other anti-HCV agents
Period: Treatment Period
Arm/Group | Treatment Naive | Treatment Experienced
Started | 54 | 24
Completed | 49 | 21
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Participant request to discontinue | 1 | 1
Not completed — Participant moved to another province | 1 | 0
Not completed — Participant was incarcerated | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Follow Up Period
Arm/Group | Treatment Naive | Treatment Experienced
Started | 50 | 23
Completed (Completed Follow-Up Period) | 50 | 21
Not Completed | 0 | 2
Not completed — Unable to return for week 24 follow-up | 0 | 1
Not completed — Unable to return for follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Naive | Treatment Experienced | Total
Number analyzed (Participants) | 54 | 24 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Treated Participants
  Years | 54 (7.97) | 55.3 (4.90) | 54.4 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Treated Participants
  Participants
    Female | 14 | 7 | 21
    Male | 40 | 17 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 20 | 8 | 28
  Unknown or Not Reported | 27 | 10 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 21 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target detected or target not detected at follow-up Week 12. HCV RNA measurements are excluded after the start of non-study anti-HCV medication on treatment or during follow-up. Modified (mITT) approach is based on treated subjects. The numerator is based on subjects meeting the response criteria and the Next Value Carried Backwards approach.
Time Frame: Week 12
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HCV Treatment Naive: HCV treatment-naive: No previous exposure to any interferon (IFN) formulation (ie, IFN or peg-IFN), RBV, or any HCV DAAs
- HCV Treatment Experienced: HCV treatment-experienced: Previous treatment with IFN/RBV, SOF + RBV, and other anti-HCV agents
Arm/Group | HCV Treatment Naive | HCV Treatment Experienced
Number analyzed (Participants) | 54 | 24
Percentage of participants | 92.6 [82.1 to 97.9] | 75.0 [53.3 to 90.2]

2. Secondary Outcome: Percentage of Participants Who Achieve SVR12 in the Presence and Absence of Baseline NS5A (Non-structural Protein 5A) Resistance-associated Polymorphisms
Description: as for outcome 1
Time Frame: Week 12 (Follow-up period)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCV Treatment Naive | HCV Treatment Experienced
Number analyzed (Participants) | 54 | 24
Percentage of participants
  NS5A-Y93 Polymorphism: YES: number analyzed (Participants) | 7 | 1
  NS5A-Y93 Polymorphism: YES | 85.7 [42.1 to 99.6] | 0.0 [0.0 to 97.5]
  NS5A-Y93 Polymorphism: NO: number analyzed (Participants) | 47 | 23
  NS5A-Y93 Polymorphism: NO | 93.6 [82.5 to 98.7] | 78.3 [56.3 to 92.5]

3. Secondary Outcome: Percentage of Subjects Who Achieve HCV RNA < LLOQ, TD or TND Through Follow up Week 24
Description: HCV RNA measurements are excluded after the start of non-study anti-HCV medication on treatment or during follow-up. Modified (mITT) approach is based on treated subjects. The numerator is based on subjects meeting the response criteria. SVR12 is based on Next Value Carried Backwards approach.
Time Frame: At Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, End of Treatment (24 weeks), Follow Up Week 4 (28 weeks), Follow Up Week 12 (36 weeks), Follow Up Week 24 (48 weeks)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | HCV Treatment Naive | HCV Treatment Experienced
Number analyzed (Participants) | 54 | 24
Percentage
  Week 1 | 14.8 [6.6 to 27.1] | 12.5 [2.7 to 32.4]
  Week 2 | 50.0 [36.1 to 63.9] | 54.2 [32.8 to 74.4]
  Week 4 | 92.6 [82.1 to 97.9] | 75.0 [53.3 to 90.2]
  Week 8 | 98.1 [90.1 to 100.0] | 91.7 [73.0 to 99.0]
  Week 12 | 92.6 [82.1 to 97.9] | 87.5 [67.6 to 97.3]
  Week 16 | 90.7 [79.7 to 96.9] | 83.3 [62.6 to 95.3]
  Week 20 | 94.4 [84.6 to 98.8] | 83.3 [62.6 to 95.3]
  Week 24 | 88.9 [77.4 to 95.8] | 87.5 [67.6 to 97.3]
  End of Treatment | 100.0 [93.4 to 100.0] | 91.7 [73.0 to 99.0]
  Follow Up Week 4 | 88.9 [77.4 to 95.8] | 79.2 [57.8 to 92.9]
  Follow Up Week 12 (Imputed) | 92.6 [82.1 to 97.9] | 75.0 [53.3 to 90.2]
  Follow Up Week 24 | 92.6 [82.1 to 97.9] | 66.7 [44.7 to 84.4]

4. Secondary Outcome: Percentage of Subjects Who Achieve HCV RNA < LLOQ, TND Through Follow up Week 24
Description: HCV RNA measurements are excluded after the start of non-study anti-HCV medication on treatment or during follow-up.
  Modified (mITT) approach is based on treated subjects. The numerator is based on subjects meeting the response criteria.
Time Frame: At Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, End of Treatment, Follow Up Week 4, Follow Up Week 12, Follow Up Week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | HCV Treatment Naive | HCV Treatment Experienced
Number analyzed (Participants) | 54 | 24
Percentage
  Week 1 | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 14.2]
  Week 2 | 11.1 [4.2 to 22.6] | 12.5 [2.7 to 32.4]
  Week 4 | 64.8 [50.6 to 77.3] | 62.5 [40.6 to 81.2]
  Week 8 | 94.4 [84.6 to 98.8] | 83.3 [62.6 to 95.3]
  Week 12 | 90.7 [79.7 to 96.9] | 83.3 [62.6 to 95.3]
  Week 16 | 90.7 [79.7 to 96.9] | 79.2 [57.8 to 92.9]
  Week 20 | 94.4 [84.6 to 98.8] | 83.3 [62.6 to 95.3]
  Week 24 | 88.9 [77.4 to 95.8] | 83.3 [62.6 to 95.3]
  End of Treatment | 100.0 [93.4 to 100.0] | 87.5 [67.6 to 97.3]
  Follow Up Week 4 | 88.9 [77.4 to 95.8] | 79.2 [57.8 to 92.9]
  Follow Up Week 12 | 90.7 [79.7 to 96.9] | 75.0 [53.3 to 90.2]
  Follow Up Week 24 | 90.7 [79.7 to 96.9] | 66.7 [44.7 to 84.4]

ADVERSE EVENTS:
Time Frame: From first dose until last dose plus 7 days (assessed up to May 2017, approximately 14 months).
Groups:
- Overall: Daclatasvir(DCV) + Sofosbuvir(SOF) + Ribavirin(RBV): Oral dosing of DCV 60 mg tablet once daily + SOF 400 mg tablet once daily + RBV 1000-1200 mg tablet per day (weight based) for 24 weeks.
Arm/Group | Overall: Daclatasvir(DCV) + Sofosbuvir(SOF) + Ribavirin(RBV) | HCV Treatment Naive | HCV Treatment Experienced
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/54 | 0/24
Serious Adverse Events (participants affected / at risk) | 8/78 | 4/54 | 4/24
Other Adverse Events (participants affected / at risk) | 63/78 | 44/54 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall: Daclatasvir(DCV) + Sofosbuvir(SOF) + Ribavirin(RBV) (N=78) | HCV Treatment Naive (N=54) | HCV Treatment Experienced (N=24)
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall: Daclatasvir(DCV) + Sofosbuvir(SOF) + Ribavirin(RBV) (N=78) | HCV Treatment Naive (N=54) | HCV Treatment Experienced (N=24)
Anaemia (Blood and lymphatic system disorders) | 10 | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 1
Nausea (Gastrointestinal disorders) | 19 | 13 | 6
Toothache (Gastrointestinal disorders) | 5 | 3 | 2
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1
Fatigue (General disorders) | 34 | 21 | 13
Nasopharyngitis (Infections and infestations) | 4 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Dizziness (Nervous system disorders) | 6 | 3 | 3
Headache (Nervous system disorders) | 22 | 14 | 8
Anxiety (Psychiatric disorders) | 5 | 3 | 2
Insomnia (Psychiatric disorders) | 14 | 11 | 3
Irritability (Psychiatric disorders) | 7 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Pyrexia (General disorders) | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 3 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 1 | 2
Oral Herpes (Infections and infestations) | 2 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 2
Pruritis Generalised (Skin and subcutaneous tissue disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02673489/SAP_000.pdf
  • Study Protocol (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02673489/Prot_001.pdf